CLINICAL TRIAL: NCT01508845
Title: A Pilot Study of the Effect of Dietary Fat Type and Amount on Vitamin D3 Absorption
Acronym: MUFA/PUFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2730
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; vitamin D absorption; vitamin D deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- High MUFA/PUFA, 1600 IU vitamin D3 (Active Comparator): Subjects will receive 3 meals (1 day) with a high MUFA/PUFA ratio (20g/5g), along with 800 IU of vitamin D3 and 800 IU of deuterated vitamin D3
  Interventions: Dietary Supplement: cholecalciferol
- High MUFA/PUFA, 50,800 IU vitamin D3 (Active Comparator): Subjects will receive 3 meals (1 day) with a high MUFA/PUFA ratio (20g/5g), along with 50,000 IU of vitamin D3 and 800 IU of deuterated vitamin D3
  Interventions: Dietary Supplement: cholecalciferol
- Low MUFA/PUFA, 50,800 IU vitamin D3 (Active Comparator): Subjects will receive 3 meals (1 day) with a low MUFA/PUFA ratio (5g/20g), along with 50,000 IU of vitamin D3 and 800 IU of deuterated vitamin D3
  Interventions: Dietary Supplement: cholecalciferol
- Fat free meal, 50,800 IU vitamin D3 (Active Comparator): Subjects will receive 3 fat-free meals (1 day) and 50,000 IU vitamin D3 and 800 IU of deuterated vitamin D3
  Interventions: Dietary Supplement: cholecalciferol

INTERVENTIONS:
Dietary Supplement: cholecalciferol — 800 IU vitamin D3, 1 dose; 800 IU deuterated vitamin D3, 1 dose
  Other Names: vitamin D3
  Arms: High MUFA/PUFA, 1600 IU vitamin D3
Dietary Supplement: cholecalciferol — 50,000 IU vitamin D3, 1 dose; 800 IU deuterated vitamin D3, 1 dose
  Other Names: vitamin D3
  Arms: High MUFA/PUFA, 50,800 IU vitamin D3
Dietary Supplement: cholecalciferol — 50,000 IU vitamin D3, 1 dose; 800 IU vitamin D3, 1 dose
  Other Names: vitamin D3
  Arms: Low MUFA/PUFA, 50,800 IU vitamin D3
Dietary Supplement: cholecalciferol — 50,000 IU vitamin D3, 1 dose; 800 IU deuterated vitamin D3, 1 dose
  Other Names: vitamin D3
  Arms: Fat free meal, 50,800 IU vitamin D3

SUMMARY:
This study will examine whether the amount and type of fat, mono-unsaturated fat (MUFA) vs. poly-unsaturated fat (PUFA), in a meal affects the absorption of vitamin D, which is taken after that meal. The study hypothesis is that vitamin D3 absorption will be greater when fat is present vs. absent in the meal. A secondary hypothesis is that vitamin D3 absorption will be greater in the presence of a meal with a high MUFA/PUFA compared with a low MUFA/PUFA ratio.

DETAILED DESCRIPTION:
There is evidence that vitamin D has a favorable effect on bone and muscle. Many adults have low blood levels of 25-hydroxyvitamin D (25OHD) and consequently, vitamin D supplements are being widely recommended. The effect of a meal on the absorption of vitamin D is poorly understood. This single blind study will examine whether the amount and type of fat in the meal with which vitamin D is taken influences its absorption. Vitamin D dissolves in fat and so dietary fat may affect its absorption; moreover the type of fat with respect to mono- and poly-unsaturation may also influence absorption. This study should increase our understanding of how best to take vitamin D in order to achieve maximal absorption. Up to 65 healthy older men and women with 25OHDlevels in the insufficient range will be enrolled in order to get 60 completers in this 1-day study. They will randomized to one of three meal groups: high MUFA/PUFA (n=30), low MUFA/PUFA (n=15), or fat-free (n=15). Those in the high MUFA/PUFA group will also be randomized to a single dose of either 1,600 or 50,800 IU of vitamin D. All participants in the other two groups will receive the 50,800 IU dose. They will consume only the three meals provided during the study day. In the morning they will come to the Center for a blood draw, to consume their breakfast meal, and to take their assigned dose of vitamin D (part of which is labeled with the non-radioactive tracer, deuterium to enable direct assessment of vitamin D absorption). They will also complete questionnaires about their diet and health and have a DXA total body scan. They will be given a boxed lunch to eat at noon. They will return to HNRCA for blood draws at 6:00, 8:00, and 10:00 pm. They will have dinner at HNRCA after the 6:00 pm blood draw. They finish the study after the final blood draw. Participants who receive the higher dose of vitamin D, 50,800 IU, will be asked not to take more than 400 IU of vitamin D or 1000 mg per day of supplemental calcium or attend tanning salons for the month after completing the study, in order to minimize any risk of symptoms from the vitamin D. Blood draws include screening visit 20 cc, morning visit 15 cc, and three evening blood draws of 15, 15, and 15 cc, respectively, total 80 cc.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men and women age 50 years and older
* Women must be at least 1 year since last menses
* Subjects must agree not to attend a tanning salon or increase their sun exposure between the screening and final study visits and, for those in the higher vitamin D dose group (50,800 IU), for one month after they have completed the study.
* Subjects must agree not to take more than 400 IU of vitamin D (the amount in most multivitamins) or 1000 mg of calcium per day as their own supplements between the screening and final study visits and, for those in the higher vitamin D dose group (50,800 IU), for one month after completing the study (Note: no supplemental calcium or vitamin D is allowed on the study day.
* Screening serum 25OHD of 25 to 29.5 ng/ml
* Screening BMI 20 to 29.5 kg/m2
* Screening plasma triglyceride concentrations below 150 mg/dL

Exclusion Criteria:

* Uncontrolled type 2 diabetes with fasting blood sugar >140 mg/dl
* GFR < 30 ml/min calculated from serum creatinine with use of the Modification of Diet in Renal Disease (MDRD) Study equation [7]
* Screening fasting spot urinary calcium:creatinine ratio (Ca:Cr) > 0.325 (corresponding to a 24-hr urine calcium of 350 mg)
* Screening serum calcium exceeding upper normal limit (reference range 8.3 -10.2 mg/dl)
* Other abnormalities in screening labs, at the discretion of the study physician (PI)
* Sarcoidosis
* Malabsorption, Crohn's disease
* Subjects with disorders of bone and mineral metabolism
* Kidney stones - in the last 3 years
* Evidence of chronic liver disease, including alcoholism
* Cancer treatment in the last year (except basal cell carcinoma) or terminal illness
* Use of lipid lowering medications, plant sterols, fish oil, or flaxseed oil
* Treatment in the last 6 months with estrogen, raloxifene, calcitonin, or testosterone (vaginal estrogen okay)
* Treatment in the last year with teriparatide or denosumab
* Treatment in the last 2 years with bisphosphonates
* Oral corticosteroid therapy for over 3 weeks within the last 6 months
* Anticonvulsant therapy
* High dose thiazide therapy (>37.5 mg per day)
* Allergy to egg
* Non-English speaking subjects (The food frequency questionnaire to be used in this study has not been validated in other languages. Thus, their diet data would not be able to be included in the analyses. As such, it is inappropriate to expose non-English speaking participants to the study risks, however small, when their data will not contribute to the study results.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The rate of vitamin D3 absorption after consuming meals with 3 different ratios of MUFA/PUFA content. | 10, 12 and 14 hours

SECONDARY OUTCOMES:
The association between changes in plasma D3 and fatty acid profiles, specifically MUFAs. | 10, 12 and 14 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bess Dawson-Hughes, M.D., Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States